CLINICAL TRIAL: NCT02330900
Title: Evaluation of Interference Between Cell Phones and Implantable Cardioverter Defibrillators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Haran Burri, MD, Dr, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-245
Record Dates: First submitted 2014-11-25; First posted 2015-01-05 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Electromagnetic Interference
Keywords: Implantable cardioverter defibrillator; Electromagnetic interference; Cell phone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (No Intervention): Evaluation of interference
  Interventions: Other: Study group

INTERVENTIONS:
Other: Study group — Exposure to cell phone interference of the ICD

SUMMARY:
Evaluation of electromagnetic interference between modern cell phones and contemporary implantable cardioverter defibrillators (ICDs)

DETAILED DESCRIPTION:
Electrograms of ICDs will be analyzed during wireless telemetry and during exposure to an activated cell phone. ICD therapy will have been temporarily inactivated before exposure to cell phones to avoid inappropriate shocks, and the sensitivity level of the ICD will be set to maximum. The cell phones will be held over the ICD generator, as well as in the parasternar region (close to the ICD lead, which senses the signals).

Interference will be assessed by the presence of visible artefacts on the real-time electrogram, with ICD marker annotations showing atrial and/or ventricular sensed episodes. The outcome measure will be the number and proportion of patients who have electromagnetic interference of the ICD when exposed to cell phones.

The procedure will take approximately 5-10minutes, with reprogramming of the device at the end of the test. No further follow-up in the context of the study will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Implantation with a wireless-enabled ICD

Exclusion Criteria:

* Age <18yrs
* inability to sign an informed consent
* pacemaker dependancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who have electromagnetic interference of the ICD when exposed to cell phones. | 5-10minutes
  Detection of electromagnetic interference

CONTACTS AND LOCATIONS:
Overall Officials: Haran Burri, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Burri H, Mondouagne Engkolo LP, Dayal N, Etemadi A, Makhlouf AM, Stettler C, Trentaz F. Low risk of electromagnetic interference between smartphones and contemporary implantable cardioverter defibrillators. Europace. 2016 May;18(5):726-31. doi: 10.1093/europace/euv374. Epub 2016 Feb 8. PMID 26857191